CLINICAL TRIAL: NCT05189990
Title: Investigation of the Electrical Impedance Tomography (EIT) Effectiveness in Detecting Fatty Liver Disease
Brief Title: Electrical Impedance Tomography in Fatty Liver Detection
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Gense Technologies Ltd. (Unknown); Innovation and Technology Commission, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Lung-Yi Mak Loey, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: HKU-DM-MAK-NAFLD01
Record Dates: First submitted 2021-12-17; First posted 2022-01-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: electrical impedance; controlled attenuation parameter; magnetic resonance imaging
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electrical impedance tomography — Fatty liver patients will be recruited from the Department of Medicine at Queen Mary Hospital. Gender- and age- matched control subjects will be publicly recruited. Subjects will undergo the EIT-liver scan and FibroScan®. Selected subgroups will also undergo MRI-PDFF scan. The performance characteristics of the device and with respect to Fibroscan/ MRI-PDFF for liver fat quantification will be assessed.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a condition where hepatocytes contain an abnormally high fat percentage. This condition is becoming increasingly common due to unhealthy food habits and sedentary lifestyle. Since NAFLD is a silent disease, many patients would be diagnosed at the advanced stages when fat accumulation, scarring and liver cell damage are irreversible. Therefore, early diagnosis of fatty liver disease during its reversible stages is warranted. Current diagnostic techniques for fatty liver disease, such as the FibroScan® and MRI proton density fat fraction (PDFF) are expensive, and require the active work of certified professionals. Electrical Impedance Tomography (EIT) is an alternative low cost, non-invasive imaging technique that does not involve radiation nor a trained operator. The electrical conductivity of biological tissues varies according to the tissue type and frequency of AC current. Fat tissue conductivity is known to be substantially stable across the EIT current injection frequency spectrum. On the other hand, liver tissue conductivity significantly increases over frequency change. Hence, the liver fat content can be measured using frequency-difference EIT (fdEIT). The aim of this study is to investigate the feasibility and effectiveness of fdEIT in detecting fatty liver. To achieve this goal, a total of 160 subjects will be recruited, paired fdEIT-Fibroscan data will be acquired. First, optimal fdEIT current injection frequency range will be determined. Second, fdEIT derived indicators will be computed and statistical analysis will be performed to verify the significance of correlation between the two. Comparative exploration between EIT and MRI-PDFF will be performed on a subset of the study population, looking at both spatial localization and image derived indicators.

Finally, demographics, clinical assessment and patient history will be analysed to produce demographic group-based insights.

DETAILED DESCRIPTION:
Fatty liver disease is a condition where the hepatocytes (liver cells) contain more than 5% fat. This condition is becoming increasingly common due to unhealthy food habits and sedentary lifestyle. Since NAFLD is a silent disease with symptoms arising only at the later stages (e.g., fibrosis), many patients would be diagnosed at the advanced stages when fat accumulation, scarring and liver cell damage are irreversible. Therefore, early diagnosis of silent fatty liver disease during its reversible stages is important to prevent cell damage, liver transplantation and allow better long-term prognosis.

Currently, liver biopsy is the gold standard in diagnosis and prognosis of fatty liver disease. However, biopsies are invasive, expensive and involve risks of internal bleeding and high sampling error. Non-invasive diagnostic tests include blood tests, FibroScan® and MRI. FibroScan® (Echosens, Paris, France) is a quick 10 minutes non-invasive test which measures the fatty change. Normal liver fat amount has controlled attenuation parameter (CAP) <248 dB/m which is S0, while mild fatty liver has CAP 248-267 dB/m or S1. Moderate fatty liver has CAP 268-279 dB/m or S2 and lastly severe fatty liver has CAP >279 dB/m or S3 (Karlas et al., 2017). The device is known to have reduced reliability for patients who are morbidly obese or have ascites. It also heavily relies on the operator experience. Another liver fat quantification method is MRI-based proton density fat fraction (MRI-PDFF). MRI-PDFF is a noninvasive imaging tool which can accurately and precisely calculate the percentage of liver fat over the whole liver. Nevertheless, MRI-PDFF takes a long time (~30 minutes), is expensive, not portable and not routinely accessible.

EIT could be an alternative low cost, noninvasive imaging technique that does not involve radiation and is routinely accessible. Existing EIT commercial devices are at present being deployed in some clinical settings. EIT technology has been in use since more than a decade, although so far it has mostly been used to assist mechanically ventilated patients in intensive care units to prevent lung damage caused by artificial ventilation.

Within the past few years, non-clinical research studies on applying EIT for fatty liver detection in animal and human models have been performed. The electrical conductivity of biological tissues varies according to the tissue type and frequency of AC current. On one hand, fat tissue conductivity is known to be substantially stable across the EIT current injection frequency spectrum. On the other hand, liver tissue conductivity significantly increases over frequency change. Hence, biological tissues can potentially be differentiated using EIT frequency spectrum analysis.

ELIGIBILITY:
Inclusion Criteria:

* Fatty liver patients diagnosed with fatty liver at S1, S2 and S3 stages, will be included.
* Control subjects will also be included (who do not have any known liver diseases). Healthy subjects will be chosen to be age and gender matched with case subjects.

Exclusion Criteria:

* Subjects with previous liver diseases (in the control group) or any liver diseases other than fatty liver (in fatty liver patients).
* Subjects who had any kind of liver surgery or liver transplantation.
* Subjects with damaged skin on the abdomen.
* Subjects with implanted electronic devices.
* Subjects with spinal diseases/discomfort
* Subjects who had any recent abdominal surgery
* Pregnant women
* Ascites
* Heavy alcohol intake
* Metallic implants

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Two populations will be included in this study:
  1. Fatty liver patients: patients diagnosed with fatty liver disease at different stages of the disease according to hepatic steatosis grade (S1-S3). These patients will be recruited from the affiliated institution of the study team.
  2. Controls: healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Optimal electrical impedance tomography (EIT) injection frequencies for fatty liver detection | 24 months
  The optimal EIT current injection frequencies used in the novel EIT-liver device for fatty liver assessment will be determined by gross data collection and fine-tuning, to shorten the EIT scan time

SECONDARY OUTCOMES:
The performance characteristics of EIT liver device in hepatic steatosis assessment compared to transient elastography | 24 months
  The correlation between the novel EIT-liver device derived data and liver stiffness obtained from transient elastography (a well-established ultrasound-based imaging for liver fat and fibrosis quantification)

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Yi Mak, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Select A State Or Province, China